CLINICAL TRIAL: NCT03605940
Title: A Multi-center Randomized Phase II Study Comparing Corticosteroids Alone Versus Corticosteroids and Extracorporal Photopheresis (ECP) as First-line Treatment of Standard Risk Grade II Acute Graft-versus-host Disease After Allogeneic Stem Cell Transplantation
Brief Title: A Study Comparing Corticosteroids Alone Versus Corticosteroids and Extracorporal Photopheresis (ECP) as First-line Treatment of Standard II Acute Graft-versus-host Disease
Acronym: PCE-aGVHD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-005162-22; PSS2017/PCE-aGVHD-RUBIO/VS (Other: CHRU Nancy)
Record Dates: First submitted 2018-07-21; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Acute-graft-versus-host Disease
Keywords: Acute-graft-versus-host Disease; Extracorporal Photopheresis
MeSH Terms: interventions — Methoxsalen; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): corticosteroids + ECP
  Interventions: Combination Product: Methoxsalen + ECP device; Drug: Corticosteroids
- Contrôl group (Active Comparator): corticosteroids alone
  Interventions: Drug: Corticosteroids

INTERVENTIONS:
Combination Product: Methoxsalen + ECP device — 2 sessions per week during 4 weeks and 1 session per week during 8 weeks
  Arms: Experimental group
Drug: Corticosteroids — 2 mg/kg/day

SUMMARY:
Acute graft versus host-disease remains a major cause of morbidity and mortality after allogeneic hematopoietic stem cell transplantation. The incidence of grade II to IV acute GVHD ranges from 30 to 50% of the patients transplanted. Steroids remain the standard first line treatment for acute GVHD.

Prolonged exposure to steroids is associated to increased risk of infections and of osteoporosis, osteonecrosis and alteration of growth in children. Thus, reducing steroid exposure in order to reduce treatment-related morbidity is another important goal in the management of standard risk aGVHD.

Extracoporeal photopheresis (ECP) is active in controlling steroid refractory or dependent acute GVHD.

Hypothesis:

In this study, the team hypothesizes that addition of ECP to first line treatment with 2 mg/kg steroids of standard risk grade II aGVHD can reduce steroid exposure by increasing the probability of 6 month FFTF including absence of systemic steroids for chronic GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years ;
* Having received an allogeneic stem cell transplantation for any malignant or non-malignant hemopathy and whatever the type of donor and graft.
* with grade II acute GVHD with skin involvement (stage 1-3 skin +/- stage 1 gastro intestinal) in the 3 months following the allogeneic stem cell transplantation
* acute GVHD in the first line treatment
* validation of the presence of peripheral or central venous access allowing to perform 2 ECP per week during 3 months. In the absence of a pre-existing and adpated central catheter at the time of inclusion, peripheral venous access will be preferred
* Leucocytes > 1.5 G/L
* Platelets > 30 G/L, Haematocrite > 27% (allowed transfusions)
* Patient affiliated to a French Social Security regimen
* information consent form signed.

Exclusion Criteria:

* acute GVHD of grade I
* acute GVHD of grade > II
* progressive hematologic disease at inclusion
* uncontrolled ongoing infection at time of inclusion: bacterial or fungal infections, increasing CMV viral load.
* patient with HIV positivity or replicative HBV or HCV infection
* Contraindications for UVADEX / photopheresis / stéroids / posaconazole / heparin
* Patient with a history of deep venous thrombosis
* Pregnancy
* Women of child bearing potentiel not using contaception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Probability of being free of treatment failure (probability of survival without relapse, additional line of treatment for aGVHD and systemic therapy for chronic GVHD) | 6 months

SECONDARY OUTCOMES:
mean of the cumulative dose of steroids | Month 1- Month 2 - Month 3 - Month 6 - Month 12
cumulative incidence rate of infections | Month 6 - Month 12
cumulative incidence of thromboembolic complications | Month 3
incidence of chronic GVHD | Month 6 - Month 12
severity of chronic GVHD | Month 6 - Month 12
incidence rate of non-relapse mortality | Month 6 - Month 12
incidence of disease relapse | Month 6 - Month 12
disease-free survival | Month 6 - Month 12
overall survival | Month 6 - Month 12
scores of health-related quality of life using the French validated FACT-BMT | Month 3 - Month 6 - Month 12
Total T cells number | Month 3 - Month 6 - Month 12
CD4 T cells number | Month 3 - Month 6 - Month 12
CD8 T cells number | Month 3 - Month 6 - Month 12
B cells number | Month 3 - Month 6 - Month 12
NK cells number | Month 3 - Month 6 - Month 12
gamma globulin number | Month 3 - Month 6 - Month 12